CLINICAL TRIAL: NCT03388684
Title: Conjoined Twins: a Report of Four Cases.
Acronym: CT
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, principal investigator, Assiut University
Other Study IDs: 17300170
Record Dates: First submitted 2017-12-25; First posted 2018-01-03 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Conjoined Twin
MeSH Terms: conditions — Twins, Conjoined

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Conjoined twin separation surgery — This study included 4 case reports on conjoined twins (CT), 2 male and three female patients; 3 of them were parasitic and one was conjoined. We operated upon 2 parasitic and one conjoined. The 1st case died preoperatively.
  Other Names: CT Separation

SUMMARY:
The present study aims to report our experience in conjoined twin separation surgery in Assuit university and pediatric hospital, Assiut university, Assiut, Egypt over a period of 20 years.

DETAILED DESCRIPTION:
A conjoined twin is a subset of monozygotic twin gestation. It's a rare phenomenon with an incidence of 1 in 50,000 to 1:100,000 births with the higher incidence in Africa and Southwest Asia. Based on the terminology proposed by Spencer and colleagues, conjoined twins are classified according to the most prominent site of conjunction into three major groups; First, twins with a ventral union; [cephalopagus (head), thoracopagus (Thorax), omphalopagus (Abdomen) and ischiopagus (pelvis)]. Second; twins with a dorsal union; [pygopagus (sacrum), rachipagus (spine, back) and craniopagus (cranium)] and lastly; twins with a lateral union that is referred to as parapagus (side). Depending on the aspect of the embryonic disc, the most common types are thoracopagus (19%).

Surgical separation of conjoined twins is extremely challenging taking in consideration the high perioperative risk. The low incidence of such surgeries and anatomical variations in each type of conjoined twins makes each separation surgery a unique experience.

ELIGIBILITY:
Inclusion Criteria:

* conjoined twins
* symmetrical or
* asymmetrical.

Exclusion Criteria:

* conjoined twins incompatible with life
* conjoined twins with decapitating medical illness.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: conjoined twins whether symmetrical or asymmetrical.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2000-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Success of the conjoined twin separation surgery | For each case was the 1 week survival
  The operative details of the separation surgery were written in details and the separation process was showen in pictures.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Professor in anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takrouney MH, Ibrahim IA, Abdel-Ghaffar HS, Abdel-Wahhab AI, Mostafa MM, Ali WN, Abd-Elaal MS. Conjoined twins: A report of four cases. Int J Surg Case Rep. 2020;73:289-293. doi: 10.1016/j.ijscr.2020.06.072. Epub 2020 Jun 20. PMID 32721891